CLINICAL TRIAL: NCT04819737
Title: Spinal Cord Lesion Detection in Multiple Sclerosis Using Novel MRI Sequences: A Pilot Study
Brief Title: Spinal Cord Lesion Detection in Multiple Sclerosis Using Novel MRI Sequences
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Freie Akademische Gesellschaft Basel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-00269; ko21Parmar
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis (MS)
Keywords: spinal cord (SC) pathology; demyelinating lesions; Spinal cord MRI; Averaged magnetization inversion recovery acquisitions (AMIRA) sequence; Swiss MS Cohort (SMSC)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Patient Health Questionnaire

STUDY DESIGN:
Intervention Model Description: All participants (embedded within the currently ongoing Swiss MS Cohort (SMSC) study) will undergo a single visit including a clinical interview, neurological examination and MRI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal Cord MRI (Experimental)
  Interventions: Procedure: SC MRI; Other: patient questionnaire

INTERVENTIONS:
Procedure: SC MRI — SC MRI (Averaged Magnetization Inversion Recovery Acquisitions (AMIRA), standard conventional SC MRI sequences, additional sequences for spinal cord MRI (sagittal-2D or 3D short tau inversion recovery, sagittal-2D or 3D phase-sensitive inversion recovery, 3D magnetization prepared 2 rapid acquisition gradient echoes (MPRAGE)). To evaluate the presences of ongoing inflammation (acute or chronic) in the SC of patients, 3D MPRAGE and 3D fluid-attenuated inversion recovery images after intravenous gadolinium (Gd) contrast administration (0.1 mmol per kg body weight) will be acquired.
Other: patient questionnaire — 12-item multiple sclerosis walking scale (MSWS-12) questionnaire: self-report measure of the impact of MS on the individual's walking ability

SUMMARY:
This study is to evaluate the sensitivity and intra-/inter-observer agreement of the averaged magnetization inversion recovery acquisitions (AMIRA) in spinal cord (SC) Multiple sclerosis (MS) lesion detection and to evaluate the additional clinical value of this sequence in clinical settings.

DETAILED DESCRIPTION:
An averaged magnetization inversion recovery acquisitions (AMIRA) sequence was proposed for SC MRI. This MR-sequence delivers excellent contrast between the SC gray and white matter as well as between the SC and cerebrospinal fluid (CSF) in clinically feasible-acquisition times. Moreover, the high quality and in-plane resolution of AMIRA images allows for segmentation of the SC gray and white matter with high accuracy and reproducibility. This study is to evaluate the sensitivity and intra-/inter-observer agreement of the averaged magnetization inversion recovery acquisitions (AMIRA) in spinal cord (SC) Multiple sclerosis (MS) lesion detection and to evaluate the additional clinical value of this sequence in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis according to established international criteria
* Steroid free period: > 4 weeks
* Participation in the Swiss MS Cohort (SMSC) study

Exclusion Criteria:

* . History of severe (other) neurological, internal or psychiatric disease with SC affection
* MRI-related exclusion criteria (questionnaire):

  1. Paramagnetic and/or superparamagnetic foreign objects in the body (especially when located close to the SC)
  2. Pacemaker
  3. Claustrophobia
  4. Pregnancy, lactation
  5. Known hypersensitivity to gadolinium-based contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of SC lesions | one time assessment (60 minutes scheduled per patient for the MRI part including preparation time outside of the scanner and actual scanning time)
  Number of SC lesions using AMIRA compared to gold-standard conventional SC MRI sequences
Inter-observer agreement on SC lesion count | one time assessment (60 minutes scheduled per patient for the MRI part including preparation time outside of the scanner and actual scanning time)
  Inter-observer agreement with regard to lesion detection using AMIRA compared to gold-standard conventional SC MRI sequences.
Presence of ongoing inflammation (acute or chronic) in the SC | one time assessment (60 minutes scheduled per patient for the MRI part including preparation time outside of the scanner and actual scanning time)
  Presence of ongoing inflammation (acute or chronic) in the SC 3D MPRAGE and 3D fluid-attenuated inversion recovery images after intravenous gadolinium (Gd) contrast administration (0.1 mmol per kg body weight)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Parmar, PD Dr. med., Principal Investigator — University Hospital Basel, Department of Neurology
Locations (1):
- University Hospital Basel, Department of Neurology, Basel, Switzerland